CLINICAL TRIAL: NCT06616389
Title: A Phase I/IIa Study of ODX (OsteoDex) in Multiple Myeloma
Brief Title: Study of ODX (OsteoDex) in Multiple Myeloma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: DexTech Medical AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ODX-MM-001
Record Dates: First submitted 2024-09-02; First posted 2024-09-27 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: Ascending dose study to evaluate safety and biological efficacy of up to 3 dose levels of ODX
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ascending dose (Other): Each subject will receive ODX treatment at 2-week intervals up to a maximum of 7 doses or until disease progression or unacceptable toxicity. The trial will consist of the following periods:
  Screening period (V0) Treatment period (V1 to V9, which includes 2 telephone contacts) Follow-up period (V10)
  The dose cohorts will be studied sequentially as follows:
  Dose cohort 1: 3.0 mg/kg ODX Dose cohort 2: 6.0 mg/kg ODX Dose cohort 3: 9.0 mg/kg ODX
  A dose escalation meeting will be called when data are available for Visit 4 of the 4th subject in a cohort. Based on the review of the safety data, the DMC will give recommendations regarding assessment of DLTs and dose escalation.
  Interventions: Drug: ODX (Osteodex)

INTERVENTIONS:
Drug: ODX (Osteodex) — Multi-center, prospective, open-label, ascending dose study to evaluate safety and biological efficacy of up to 3 dose levels of ODX.

SUMMARY:
The current phase I/IIa trial is a multi-center, prospective, open-label, ascending dose study to evaluate safety and biological efficacy of up to 3 dose levels of ODX. Each dose cohort will consist of 4 subjects. Each subject will receive up to 7 doses of ODX, given at 2-week intervals, until unacceptable toxicity or disease progression. A follow-up visit will be conducted 2 weeks after the last dose.

Primary objectives:

• To determine the safety and tolerability of ODX in subjects with relapsed/refractory multiple myeloma.

Secondary objectives:

* To evaluate the preliminary efficacy of ODX, as determined by the IMWG response criteria, in subjects with relapsed/refractory multiple myeloma.
* To evaluate the efficacy of ODX on serum biomarkers (M-protein, FLC, CTX, osteocalcin, and bone-specific S-ALP) in subjects with relapsed/refractory multiple myeloma.

Exploratory objective

• To evaluate time to progression by following M-protein and FLC levels as per clinical routine

ELIGIBILITY:
Inclusion Criteria:

* 1. Subject (male or female) is ≥ 18 years of age at the time of signing the informed consent form (ICF).

  2. Documented diagnosis av multiple myeloma according to the International Myeloma Working Group (IMWG) diagnostic criteria.

  3. Measurable disease defined as either:
  * Serum monoclonal paraprotein (M-protein) level ≥ 0.5 g/dL or urine M-protein level ≥ 200 mg/24 hours; or
  * Light chain multiple myeloma without measurable disease in the serum or the urine: Serum immunoglobulin free light chain (FLC) ≥ 10 mg/dL and abnormal serum immunoglobulin kappa lambda FLC ratio.

    4. Subjects must have received 1-5 prior lines of therapy including a PI, IMiD and CD38 antibody*.

    *Patients eligible for inclusion should have received said treatments, i.e., according to clinical routine, unless contraindicated due to induced morbidity.

    5. Subjects must have documented evidence of progressive disease based on the IMWG criteria on or after their last line of therapy.

    6. Performance status ECOG 0-2 7. Laboratory requirements:

Haematology:

Neutrophils ≥ 1.0 x 109/l Hemoglobin ≥ 80 g/l Platelets ≥ 50 x 109/l

Hepatic function:

Total S/P-bilirubin ≤ 1.5 times the upper limit of normal (ULN) AST (SGOT) / ALT (SGPT) ≤ 2.5 times ULN

Renal function:

S/P-creatinine ≤ 1.5 times ULN

Electrolytes:

S/P-sodium, S/P-potassium, S/P-calcium corrected for S/P albumin , S/P-phosphate, and S/P magnesium, all within normal ranges. At the discretion of the Investigator, supplements may be given to correct these values, in which case electrolytes must be shown to be within normal ranges before inclusion into the study.

8. No evidence (< 5 years) of prior malignancies (except successfully treated basal cell or squamous cell carcinoma of the skin).

9. Able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

1. Concurrent use of other anti-cancer agents/treatments.
2. Any treatment modalities involving chemotherapy, radiation, or major surgery within 4 weeks prior to treatment in this study.
3. Simultaneous participation in any other study involving investigational drugs or having participated in an investigational study less than 4 weeks prior to start of study treatment.
4. Any condition, including the presence of laboratory abnormalities, which confounds the ability to interpret data from the study or places the patient at unacceptable risk if he or she participates in the study.
5. Known active CNS involvement or exhibits clinical signs of meningeal involvement of multiple myeloma.
6. Plasma cell leukemia, Waldenstrom's macroglobulinemia or POEMS syndrome.
7. Dental surgery (dental extraction), periodontal disease, local trauma including poorly fitting dentures within 6 months prior to the first dose of study drug.
8. Treatment with bisphosphonates or denosumab within 6 weeks prior to first dose of study medication.
9. Male subjects not willing to use condom to prevent pregnancy and drug exposure of a fertile female partner and refrain from donating sperm from the date of the first dose until the end of study treatment.
10. Pregnant or breastfeeding females.
11. Female subjects of childbearing potential** not willing to use a contraceptive method with a failure rate of < 1% to prevent pregnancy during study treatment. Highly effective birth control methods include:

    * combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation:

      * oral
      * intravaginal
      * transdermal
    * progestogen-only hormonal contraception associated with inhibition of ovulation:

      * oral
      * injectable
      * implantable
    * intrauterine device
    * intrauterine hormone-releasing system (for example, progestin-releasing coil)
    * vasectomized male (with appropriate post vasectomy documentation of the absence of sperm in the ejaculate)
    * bilateral tubal occlusion or hysterectomy. **Female subjects are considered of non-childbearing potential if they are pre-menopausal females with a documented tubal ligation or hysterectomy or bilateral oophorectomy; or as post-menopausal females defined as at least 12 months of amenorrhea.
12. Subjects in which pre-medication with dexamethasone, antihistamine, and paracetamol would be contraindicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-11-29 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
To determine the incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] in subjects with relapsed/refractory multiple myeloma myeloma. | During the 14 week treatment/follow up period
  Number of participants with AEs/SAEs, with abnormal vital signs, abnormal physical examination findings, abnormal ECG readings, and abnormal results of urinalysis and safety laboratory tests (haematology, electrolytes, liver function, and biochemistry including S/P-Creatinine and S/P-Cystatin C)

SECONDARY OUTCOMES:
To evaluate the preliminary efficacy of ODX, as determined by the IMWG response criteria, in subjects with relapsed/refractory multiple myeloma. | During the 14 week treatment/follow up period
  Best overall response rate (partial response [PR] or better) reached during the 14-week treatment/follow-up period, as measured by the IMWG response criteria.
To evaluate the efficacy of ODX on serum biomarkers (M-protein, FLC, CTX, osteocalcin, and bone-specific S-ALP) in subjects with relapsed/refractory multiple myeloma. | During the 14 week treatment/follow up period
  Change in the levels of the serum biomarkers M-protein, FLC, CTX, osteocalcin, and bone-specific S ALP from baseline to Weeks 2, 4, 6, 8, 10, 12, and 14.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Holmberg, Study Chair — DexTech Medical AB
Locations (2):
- Sweden (2):
  - Karolinska Universitetssjukhuset Huddinge Cancerstudieenheten M62, Stockholm
  - Uddevalla Sjukhus, Hematologens dagvård, Uddevalla

IPD SHARING:
Plan to Share IPD: No